CLINICAL TRIAL: NCT01458808
Title: Effects of Dietary and Dialysate Sodium Reduction on Body Fluid Volume and Inflammatory State in Hemodialysis Patients. A Prospective Randomized Controlled Study
Brief Title: Dietary and Dialysate Sodium Reduction on Body Fluid Volume and Inflammatory State in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Principal Investigator, Lidiane Silva RodriguesTelini, MSC, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-55
Record Dates: First submitted 2011-06-14; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Kidney Diseases Stage 5
Keywords: salt; inflammation; hypervolemia; diet
MeSH Terms: conditions — Inflammation; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Composed by 21 patients treated with reduction of 2 grams of sodium reduction in their habitual diet.
  Interventions: Other: Dietary sodium restriction
- Group B (Experimental): Composed by 20 patients treated by reduction of dialysate concentration from 138 to 135 mEq/L
  Interventions: Other: Dialysate sodium concentration reduction
- Group C (No Intervention): Composed by 18 patients followed without changes in dialysate sodium concentration or diet sodium amount.

INTERVENTIONS:
Other: Dietary sodium restriction — Restriction of 2 grams on daily sodium diet intake.
  Other Names: Dietary prescription
  Arms: Group A
Other: Dialysate sodium concentration reduction — Reduction of dialysate sodium concentration from 138 to 135 mEq/L
  Other Names: Dialysis prescription
  Arms: Group B

SUMMARY:
Objective: To evaluate the influence of dietary sodium reduction on body fluid volume and inflammatory state in hemodialysis (HD) patients.

Design: Prospective controlled randomized study. Setting: Dialysis Unit of Botucatu Medical School Hospital, Sao Paulo State University, Brazil.

Patients: Adult patients on HD for at least 30 days and C-reactive protein (CRP) ≥ 0.7 mg/dl were randomly allocated into two groups: Group A: 21 patients treated with a 2g sodium restriction in their habitual diet, and Group B: 18 controls. Inflammatory, biochemical, hematological and nutritional markers, as well as dialysis dosage were assessed at baseline and after 8 and 16 weeks.

DETAILED DESCRIPTION:
The prognosis of chronic kidney diseases (CKD) patients is strongly compromised by cardiovascular (CV) complications. Inflammation is established as a major risk factor for CV complications in these patients, occurring in approximately one third of them. Recently, growing evidences have suggested the body water volume expansion is a cause of inflammation in CKD. In a previous study Rodrigues Telini showed that dietary sodium restriction reduced the inflammatory markers levels in hemodialysis (HD) patients. Similar results were observed in patients treated by reduction of HD dialysate sodium concentration. However in both studies no significant reduction in body volume markers was observed. These results could be due to small number of patients or low sensibility of volume markers; on the other hand they could suggest a direct role of sodium as an inflammatory inducer independently of volume. With a larger number of patients and using a more sensitive volume marker as the B-type natriuretic peptide (BNP), this study intends to confirm the hypothesis that sodium mobilization can reduce the body water volume and attenuate the inflammatory in HD patients. A hundred thirty-five patients will be enrolled and divided in three groups with 35 patients: A, treated by reduction of 2 grams in daily sodium intake; B, exposed to reduction of sodium dialysate from 138 to 135 mEq/L and C, control group. The patients will be followed up by 16 weeks and inflammatory markers (CRP, interleukin-6, and tumor necrosis factor) as well as volume markers (Watson formula, electrical bioimpedance measurements and BNP concentration) will be determine each 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* included patients aged ≥ 18 years who had been on hemodialysis for at least 90 days, and were diagnosed with inflammation. Inflammation was defined as C Reactive Protein ≥ 0.7 mg/dL

Exclusion Criteria:

* acute inflammatory processes confirmed by clinical criteria and/or complementary tests
* acute inflammatory diseases
* tuberculosis
* use of antibiotics within the past two months
* chronic inflammatory diseases
* neoplasias
* chronic obstructive pulmonary disease
* use of central venous catheter and positive HIV serology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | up to 16 weeks
  The outcome will be evaluates each eight weeks
interleukin-6 | up to 16 weeks
  The outcome will be evaluates each eight weeks
alpha tumor necrosis serum concetrations | up to 16 weeks
  The outcome will be evaluates each eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lidiane R. Telini, MSC, Principal Investigator — UPECLIN HC FM Botucatu Unesp

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803